CLINICAL TRIAL: NCT06028789
Title: Differential Diagnosis of Sterile Systemic Inflammation and Sepsis in Patients Undergoing Thoracic Aortic Surgery
Brief Title: AOrtic Surgery: Systemic Inflammatory Response Versus Sepsis
Acronym: AOSIS
Status: Recruiting | Type: Observational
Sponsor: University Hospital Hradec Kralove (Other)
Collaborators: American Association for Thoracic Surgery (Unknown)
Responsible Party: Sponsor
Other Study IDs: 202202 P02
Record Dates: First submitted 2023-05-22; First posted 2023-09-08 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Systemic Inflammatory Response Syndrome; Infections; Thoracic Aortic Aneurysm; Aortic Diseases; Immunological Abnormality
Keywords: systemic inflammatory response syndrome; infection; thoracic aortic surgery
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome; Infections; Aortic Aneurysm, Thoracic; Aortic Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Patients undergoing elective thoracic aortic surgery.
  Interventions: Diagnostic Test: Blood sample test; Procedure: Thoracic Aortic Surgery
- Control group: Patients admitted to our institution with active infectious endocarditis.
  Interventions: Diagnostic Test: Blood sample test

INTERVENTIONS:
Diagnostic Test: Blood sample test — The following groups of biomarkers will be examined:
  * standard panel of inflammation markers: CRP, PCT, IL-6, Leukocyte count, differential blood count
  * microbiology cultures according to the clinical status
  * serum biomarkers: sCD64, sTREM-1, calprotectin, pentraxin 3
  * flow cytometry: HLA-DR, CD14, CD16, CD40, CD45, CD64, CD163 expression on granulocytes and monocytes
  * cell function assay: IL-18 and IFN-γ
  * hematology: ICIS, Neutrophil-to-lymphocyte ratio - examined together with conventional hematological parameters.
  The schedule of blood sample taking will be as follows:
  A. the study group: preoperatively (T-1), 1st postoperative day (T1), 3rd postoperative day (T2), 7th postoperative day (T3), 10th postoperative day (T4)
  B. the control group: at admission or the next day (T1), 3rd day of hospital stay (T2), 7th day of hospital stay (T3), 10th day of hospital stay (T4)
Procedure: Thoracic Aortic Surgery — Scheduled surgical intervention, i.e. replacement of pre-specified part of thoracic aorta by a vascular prosthesis.
  Groups: Study group

SUMMARY:
The goal of the prospective observational study is to evaluate the immunological background of inflammatory response often seen after open thoracic aortic surgery. Patients scheduled for this type of procedure will undergo a series of blood testing (preoperatively, and several times postoperatively). The blood samples will be used for a wide scale of immunological tests to better evaluate potential differential markers against infection. A control group will include patients with active infective endocarditis (preoperatively).

The main question is if there is a biomarker able to determine a difference between sterile systemic inflammation and infection after thoracic aortic surgery. The second question is if there is a difference in dynamics of evaluated biomarkers between sterile postoperative inflammation and active endocarditis.

DETAILED DESCRIPTION:
It has been observed in daily clinical practice that patients after thoracic aortic replacement (of any extent, of any reason) often develop a set of specific symptoms. Those include fever, weakness and prolonged rise of standard laboratory parameters of inflammation (CRP and leucocyte level) in absence of infection. Those symptoms may, but do not have to, coincide with typical signs of postcardiotomy syndrome, rather characteristic by pericardial / pleural effusion and indifferent chest pain. They rather resemble a so called "postimplantation" syndrome, described after endovascular aortic repair. As a reaction to foreign vascular graft material, pro-inflammatory cytokines are being released, thus leading to flu-like symptoms in absence of true infection. Those occur in the short-term postoperatively, usually in the first 2 weeks after the surgery.

Patients after thoracic aortic surgery represent a high-risk patient cohort vulnerable to infections of any kind, mostly respiratory, urinary, wound infections, and, last but not least, early valve endocarditis / endoaortitis being the most feared of them. While clinicians (and patients) are often afraid of the abovementioned complications, the patients are forced to undergo complex diagnostic process including repeated echocardiography, collection of microbiology cultures and blood samples, chest computer tomography imaging with extensive radiation burden. The prolonged broad-spectrum empiric antibiotic treatment is often in place together with prolonged hospital stay and limited patient satisfaction. The question of starting the immunosuppressive treatment is often weighed against the potential aggravation of infection with eventual fatal consequences.

In absence of a specific biomarker to distinguish between the sterile systemic inflammation and infection, the clinicians must rely on complex evaluation of patient symptoms, clinical examination, imaging modalities, standard laboratory measures of inflammation and microbiology cultures (with some delay). However, in the era of molecular biology and extensive progress in immunology research, there has been a long row of potential biomarkers able to specify the etiology of inflammatory process significantly sooner.

The potential biomarkers of inflammation suitable for this issue are mentioned in detail further. Conventional biomarkers include CRP, leukocyte count, differential blood count, recently also procalcitonin (PCT), tumor necrosis factor-α (TNF- α) and interleukin-6 (IL-6). Hematology tests have reported novel early markers of sepsis, e.g. mean neutrophil volume or neutrophil-to-lymphocyte ratio. Novel serology markers (mostly assessed by ELISA) include soluble triggering receptor expressed on myeloid cell-1 (sTREM-1), presepsin, serum amyloid-A, pentraxin 3, hemoxygenase-1 (HO-1), soluble CD64 (sCD64), soluble CD163 (sCD163), high mobility group box-1 (HMGB-1), lipopolysaccharide-binding protein (LBP) and others. Newly, the molecules expressed on the surface of circulating blood cells may be examined using flow cytometry: CD64 on polymorphonuclears (PMN CD64 index) or monocytes, CD163, CD167, HLA-DR etc. Cell function assays which test ability of blood cells to respond to microbial stimuli (represented by LPS, flagellin, etc.) may reveal changes in soluble biomarkers, such as IL-18 or IFN-γ that reflect nature of inflammation in patients.

Recently, several scoring systems have emerged combining panels of various biomarkers. There is a promising evidence for a composite of serum and cell-expressed parameters, called "Bioscore", including procalcitonin, sTREM-1 and PMN CD64 index. A composite of 5 hematological parameters has proven to be a reliable marker of early sepsis, being called intensive care infection score (ICIS). Another scoring systems have been developed by group of Kofoed et al. Nevertheless, most of these scoring systems have been tested in the settings of unstable patients in the intensive care unit. The issue of inflammatory response described above is mostly a matter of stable patients in the standard ward who develop signs of undetermined inflammation. Eventual diagnostic modalities in these settings have been only scarcely evaluated before. The topic of inflammatory response after aortic surgery (IRAS) has not been studied in the literature yet.

ELIGIBILITY:
Inclusion Criteria (for study group):

* patient scheduled for elective replacement of thoracic aorta of any extent by artificial vascular graft, including Bentall procedure, Yacoub procedure, supracoronary aortic replacement, also Ross procedure with supracoronary aortic replacement, hemiarch and total aortic arch replacement
* signature of informed patient consent

Exclusion Criteria (for study group):

* active endocarditis or other infection
* unstable preoperative condition

Inclusion Criteria (for control group):

* patient with active infectious endocarditis
* signature of informed patient consent

Exclusion Criteria (for control group):

* more than 5 days since diagnosis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study group is defined as patients scheduled for elective replacement of thoracic aorta of any extent by artificial vascular graft, including Bentall procedure,valve-sparing root replacement, supracoronary aortic replacement, also Ross procedure with supracoronary aortic replacement, hemiarch and total aortic arch replacement.
  Control group is defined as patients admitted to our institution with active infectious endocarditis.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Serum concentration of sCD64 | After completion of the study - until the end of 2023
  A statistically significant difference in absolute value or dynamics of serum concentrations of sCD64 between the study groups to help distinguish between the specified clinical syndromes.
Expression of CD64 on granulocytes | After completion of the study - until the end of 2023
  A statistically significant difference in absolute values or dynamics of the expression of CD64 on granulocytes between the study groups to distinguish between the specified clinical syndromes. Expression on monocytes will be also assessed.
Cell function assay of INF-γ | After completion of the study - until the end of 2023
  A significant difference in the outcomes of cell function assay of INF-γ between the study groups to distinguish between the specified clinical syndromes.

SECONDARY OUTCOMES:
Serum concentration of sTREM-1 | After completion of the study - until the end of 2023
  A statistically significant difference in absolute value or dynamics of serum concentrations of sTREM-1 between the study groups to help distinguish between the specified clinical syndromes.
Serum concentration of calprotectin | After completion of the study - until the end of 2023
  A statistically significant difference in absolute value or dynamics of serum concentrations of calprotectin between the study groups to help distinguish between the specified clinical syndromes.
Serum concentration of pentraxin 3 | After completion of the study - until the end of 2023
  A statistically significant difference in absolute value or dynamics of serum concentrations of pentraxin 3 between the study groups to help distinguish between the specified clinical syndromes.
Expression of HLA-DR on granulocytes | After completion of the study - until the end of 2023
  A statistically significant difference in absolute values or dynamics of the expression of HLA-DR on granulocytes between the study groups to distinguish between the specified clinical syndromes. Expression on monocytes will be also assessed.
Expression of CD-14 on granulocytes | After completion of the study - until the end of 2023
  A statistically significant difference in absolute values or dynamics of the expression of CD-14 on granulocytes between the study groups to distinguish between the specified clinical syndromes. Expression on monocytes will be also assessed.
Expression of CD-16 on granulocytes | After completion of the study - until the end of 2023
  A statistically significant difference in absolute values or dynamics of the expression of CD-16 on granulocytes between the study groups to distinguish between the specified clinical syndromes. Expression on monocytes will be also assessed.
Expression of CD-40 on granulocytes | After completion of the study - until the end of 2023
  A statistically significant difference in absolute values or dynamics of the expression of CD-40 on granulocytes between the study groups to distinguish between the specified clinical syndromes. Expression on monocytes will be also assessed.
Expression of CD-45 on granulocytes | After completion of the study - until the end of 2023
  A statistically significant difference in absolute values or dynamics of the expression of CD-45 on granulocytes between the study groups to distinguish between the specified clinical syndromes. Expression on monocytes will be also assessed.
Expression of CD-163 on granulocytes | After completion of the study - until the end of 2023
  A statistically significant difference in absolute values or dynamics of the expression of CD-163 on granulocytes between the study groups to distinguish between the specified clinical syndromes. Expression on monocytes will be also assessed.
Cell function assay of IL-18 | After completion of the study - until the end of 2023
  A significant difference in the outcomes of cell function assay of IL-18 between the study groups to distinguish between the specified clinical syndromes.
ICIS score | After completion of the study - until the end of 2023
  A significant difference in the absolute values or dynamics of ICIS (intensive care infection score) score value between the study groups.

OTHER OUTCOMES:
Serum concentration of C-Reactive protein | After completion of the study - until the end of 2023
  A significant difference in the absolute values or dynamics of C-Reactive protein serum concentrations value between the study groups.
Serum concentration of procalcitonin | After completion of the study - until the end of 2023
  A significant difference in the absolute values or dynamics of procalcitonin serum concentrations value between the study groups.
Serum concentration of IL-6 | After completion of the study - until the end of 2023
  A significant difference in the absolute values or dynamics of IL-6 serum concentrations value between the study groups.
Leukocyte blood count | After completion of the study - until the end of 2023
  A significant difference in the absolute values or dynamics of leukocyte blood count values between the study groups. Differential blood count will also be included in analysis.
Neutrophil-to-lymphocyte ratio | After completion of the study - until the end of 2023
  A significant difference in the absolute values or dynamics of neutrophil-to-lymphocyte values between the study groups.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Vojacek, Prof. MD, Study Chair — University Hospital Hradec Kralove
Locations (1):
- University Hospital Hradec Králové, Hradec Králové, Královehradecký Kraj, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gabaldo K, Sutlic Z, Miskovic D, Knezevic Pravecek M, Prvulovic D, Vujeva B, Cvitkusic Lukenda K, Hadzibegovic I. Postpericardiotomy syndrome incidence, diagnostic and treatment strategies: experience AT two collaborative centers. Acta Clin Croat. 2019 Mar;58(1):57-62. doi: 10.20471/acc.2019.58.01.08. PMID 31363326
- [Background] Daye D, Walker TG. Complications of endovascular aneurysm repair of the thoracic and abdominal aorta: evaluation and management. Cardiovasc Diagn Ther. 2018 Apr;8(Suppl 1):S138-S156. doi: 10.21037/cdt.2017.09.17. PMID 29850426
- [Background] Raveendran AV, Kumar A, Gangadharan S. Biomarkers and newer laboratory investigations in the diagnosis of sepsis. J R Coll Physicians Edinb. 2019 Sep;49(3):207-216. doi: 10.4997/JRCPE.2019.308. PMID 31497788
- [Background] Gibot S, Bene MC, Noel R, Massin F, Guy J, Cravoisy A, Barraud D, De Carvalho Bittencourt M, Quenot JP, Bollaert PE, Faure G, Charles PE. Combination biomarkers to diagnose sepsis in the critically ill patient. Am J Respir Crit Care Med. 2012 Jul 1;186(1):65-71. doi: 10.1164/rccm.201201-0037OC. Epub 2012 Apr 26. PMID 22538802
- [Background] Nierhaus A, Linssen J, Wichmann D, Braune S, Kluge S. Use of a weighted, automated analysis of the differential blood count to differentiate sepsis from non-infectious systemic inflammation: the intensive care infection score (ICIS). Inflamm Allergy Drug Targets. 2012 Apr;11(2):109-15. doi: 10.2174/187152812800392841. PMID 22280231
- [Background] Kofoed K, Andersen O, Kronborg G, Tvede M, Petersen J, Eugen-Olsen J, Larsen K. Use of plasma C-reactive protein, procalcitonin, neutrophils, macrophage migration inhibitory factor, soluble urokinase-type plasminogen activator receptor, and soluble triggering receptor expressed on myeloid cells-1 in combination to diagnose infections: a prospective study. Crit Care. 2007;11(2):R38. doi: 10.1186/cc5723. PMID 17362525
- [Background] Djebara S, Biston P, Fosse E, Daper A, Joris M, Boudjeltia KZ, Lelubre C, Cauchie P, Piagnerelli M. Time Course of CD64, a Leukocyte Activation Marker, During Cardiopulmonary Bypass Surgery. Shock. 2017 Feb;47(2):158-164. doi: 10.1097/SHK.0000000000000751. PMID 27648690
- [Background] Kolackova M, Kudlova M, Kunes P, Lonsky V, Mandak J, Andrys C, Jankovicova K, Krejsek J. Early expression of FcgammaRI (CD64) on monocytes of cardiac surgical patients and higher density of monocyte anti-inflammatory scavenger CD163 receptor in "on-pump" patients. Mediators Inflamm. 2008;2008:235461. doi: 10.1155/2008/235461. PMID 18320015